CLINICAL TRIAL: NCT07210606
Title: Central Apnea in Heart Failure: Physiological Mechanisms to Inform Treatment
Acronym: CSA-HF
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NURR-010-25S; 2I01RD001576-07A1 (Other Grant/Funding Number: CSR&D)
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Sleep Disordered Breathing; Able Bodied
Keywords: Central Sleep Apnea; Polysomnography (PSG); Respiratory Arousal Threshold; Apnea Hypopnea Index; Central Apnea Hypopnea Index; Breathing Instability; Apneic Threshold (AT); Peripheral Chemoreflex Sensitivity; CO2 reserve; Plant gain; Controller gain; Cheyne Stokes Breathing (CSB); Carotid Body Function; Peripheral Chemoresponsiveness; Heart Failure
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Central; Cheyne-Stokes Respiration; Heart Failure | interventions — Trazodone; Oxygen

STUDY DESIGN:
Intervention Model Description: Specific Aim (1) is to determine the effect of decreasing respiratory arousals on the propensity to CSA. The investigators hypothesize that combined therapy with PAP and trazodone will be superior to PAP alone in elevating the arousal threshold, widening the CO2 reserve, and decreasing CSA indices. Specific Aim (2) is to determine the effect of decreased peripheral chemoreceptor sensitivity on the propensity to CSA. The investigators hypothesize that combined therapy with PAP and supplemental O2 will be superior to PAP alone in widening the CO2 reserve, reducing controller gain, and decreasing CSA indices.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trazodone (Active Comparator): To determine the effect of dampening respiratory arousals. The investigators hypothesize that PAP therapy with trazodone at 100 mg will be superior to CPAP alone in widening the CO2 reserve during sleep, decreasing respiratory arousals, and increasing the arousal threshold.
  Interventions: Drug: Trazodone + PAP therapy
- Oxygen (Active Comparator): To determine the effect of dampening peripheral chemoreceptor sensitivity. The investigators hypothesize that supplemental oxygen will be superior to CPAP alone in widening the CO2 reserve during sleep. The secondary analysis will use CAI as supplemental oxygen, which may obscure the detection of hypopneas based on desaturation.
  Interventions: Drug: Oxygen + PAP therapy

INTERVENTIONS:
Drug: Trazodone + PAP therapy — The central apnea index and the apneic threshold will be compared under two conditions: trazodone or placebo. In addition, participants will get PAP therapy during both the conditions.
  Arms: Trazodone
Drug: Oxygen + PAP therapy — The central apnea index and the apneic threshold will be compared under two conditions: oxygen or room air. In addition, participants will get PAP therapy during both the conditions.
  Arms: Oxygen

SUMMARY:
Central sleep apnea (CSA) is common in patients with heart failure and those using opioid analgesics. Unfortunately, effective treatment of central apnea remains elusive, pressure therapy given the modest efficiency of positive airway pressure therapy. The focus of this proposal is to identify mechanistic pathways to guide future therapeutic interventions for central sleep apnea based on the strong premise that multi-modality therapy will normalize respiration and hence mitigate adverse long-term consequences of CSA. The investigators' proposed studies will test combination therapies, including positive airway pressure (PAP) plus a pharmacological agent who have heart failure or are using opioid analgesics. The investigators anticipate that findings will inform future clinical trials to improve care and quality of life among Veterans suffering from central sleep apnea, which remains difficult to treat using existing approaches.

DETAILED DESCRIPTION:
The objective in this project is to test mechanistic pathways to inform future clinical studies investigating the potential treatment of central sleep apnea (CSA) in Veterans with heart failure and reduced ejection fraction (HF). The long-term goal is to transform the care of Veterans living with these two conditions. The investigators will test two key determinants of recurrent CSA in Veterans with HF: augmented peripheral chemoreceptor activity and respiratory arousals. Specifically, the project will utilize a novel PAP plus approach, combining PAP therapy to alleviate upper airway obstruction with a specific intervention to target the mechanistic underpinnings of CSA. The experiments will capitalize on the plasticity of the CO2 reserve as the gateway to the resolution of CSA. The investigators will suppress arousals or dampen augmented PCR activity while maintaining upper airway patency with PAP. The long-term goal is to inform future multi-modality intervention studies. To this end, the following Specific Aims will be addressed in Veterans with HF and CSA. Specific Aim (1): To determine the effect of decreasing respiratory arousals on the propensity to CSA. The investigators hypothesize that combined PAP and trazodone therapy will be superior to PAP alone in elevating the arousal threshold, widening the CO2 reserve (primary outcome), and decreasing CSA indices. Specific Aim (2): To determine the effect of decreased peripheral chemoreceptor sensitivity on the propensity to CSA. The investigators hypothesize that combined PAP and supplemental O2 (targeting peripheral chemoreceptor sensitivity) will be superior to PAP alone in widening the CO2 reserve (primary outcome), reducing controller gain, and decreasing CSA indices. The proposed studies are innovative, testing mechanistic "PAP Plus" approach targeting underlying causes of CSA and alleviating upper airway obstruction with PAP. These studies will inform future clinical trials to transform central apnea care in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women Veterans with central sleep apnea, defined as Apnea Hypopnea Index (AHI)>15/hour with CAHI>5/hour, will be included with the experiments.
* Those with chronic, stable heart failure with reduced ejection fraction, receiving stable optimized guideline-based therapy and no hospitalizations or change in the medical regimen for the past 90 days before enrollment.

Exclusion Criteria:

* less than 18 years old
* pregnant or breastfeeding females
* moderate or severe obstructive or restrictive lung disease, including supplemental o2 use
* current treatment for CSA, including any form of PAP in the past three months, or phrenic nerve situation.
* too ill to engage in the study procedures, inability to provide consent for participation.
* a history of cardiac arrhythmia
* Alcohol or substance abuse (less than 90 days sobriety) or current participation in a treatment program
* depression or a history of suicidality
* severe insomnia (ISI>21) or reported short sleep duration (<6 hours)
* PAP-emergent central sleep apnea
* Lack of PAP acceptance/adherence after a one-week home PAP trial after enrollment.

Additional Trazodone Exclusions:

* Prolonged QT on baseline ECG, using medications that inhibit CYP3A4
* Patients with severe renal impairment (GFR < 20ml/min/1.73m2) or end-stage renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
CO2 Reserve | 120 days
  CO2 reserve is the requisite change to induce central apnea to as the CO2 reserve, which can be positive or negative.

SECONDARY OUTCOMES:
Peripheral Chemoresponsiveness | 120 days
  Peripheral chemoreflex sensitivity/Peripheral chemoresponsiveness is measured either via brief hypoxia or a single breath of CO2.
Arousal Threshold | 120 days
  Arousal threshold is a measure of the upper airway muscle response to an obstructive sleep event.
Carotid body function | 120 days
  This measure represents the activity of the carotid bodies. It is measured by the decrease in ventilation in response to a single breath of 100% oxygen.
Controller gain | 120 days
  Controller gain is a ventilatory response to changes in end-tidal PCO2.
Plant gain | 120 days
  Plant gain is blood gas response to a change in ventilation. This measure represents the effectiveness of the "plant" in eliminating CO2.

CONTACTS AND LOCATIONS:
Overall Officials: M Safwan Badr, MD, Principal Investigator — John D. Dingell VA Medical Center, Detroit, MI
Locations (1):
- John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No